CLINICAL TRIAL: NCT00769041
Title: A Blinded, Randomized Crossover Trial to Define the ECG Effects of TA-1790 (Avanafil) Using a Single Clinical and a Supratherapeutic Dose Compared to Placebo and Moxifloxacin in Healthy Men: A Thorough ECG Trial
Brief Title: A Thorough EKG Safety Study of TA-1790 (Avanafil)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: VIVUS LLC (Industry)
Collaborators: Covance (Industry)
Responsible Party: Wesley Day, VP Clinical, VIvus, Inc.
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: TA-140
Record Dates: First submitted 2008-10-06; First posted 2008-10-08 (Estimated); Last update posted 2011-01-07 (Estimated); Status verified 2011-01

CONDITIONS: Erectile Dysfunction
MeSH Terms: conditions — Erectile Dysfunction | interventions — Moxifloxacin; avanafil; Sugars

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- placebo (Placebo Comparator)
  Interventions: Drug: sugar pill
- moxifloxacin (Active Comparator)
  Interventions: Drug: moxifloxacin
- avanafil therapeutic (Experimental): avanafil 100mg - therapeutic dose
  Interventions: Drug: avanafil
- avanafil supratherapeutic (Experimental): avanafil 800mg - supratherapeutic dose
  Interventions: Drug: avanafil

INTERVENTIONS:
Drug: moxifloxacin — 400mg
  Arms: moxifloxacin
Drug: avanafil — 100mg single dose
  Arms: avanafil therapeutic
Drug: avanafil — 800mg single dose
  Arms: avanafil supratherapeutic
Drug: sugar pill — single dose
  Arms: placebo

SUMMARY:
This study is to assess whether treatment with a therapeutic (100 mg) or supratherapeutic (800 mg) dose of avanafil has the potential to cause QT/QTc prolongation in healthy volunteers.

ELIGIBILITY:
Inclusion Criteria:

1. Male;
2. Between 18 and 45 years of age, inclusive;
3. Have a BMI ranging between 19 and 28 kg/m2, inclusive;
4. Have no clinically significant abnormal findings on the physical examination, ECG, blood pressure, HR, medical history, or clinical laboratory results during Screening;
5. Be willing and able to comply with all trial requirements; and
6. Have given written informed consent.

Exclusion Criteria:

1. Subjects who have participated in another clinical trial of an within the last 30 days or are currently participating in another trial of an investigational drug.
2. Subjects who have participated in a previous clinical trial with avanafil.
3. Subjects who have a known allergy or hypersensitivity to avanafil, sildenafil (ViagraÂ®), vardenafil (LevitraÂ®), tadalafil (CialisÂ®) or any of the components of these drug products; moxifloxacin or its components; or to any quinolone antibiotic.
4. Subjects who have experienced dose-limiting adverse effects during therapy with a PDE5
5. Subjects who have any condition possibly affecting drug absorption
6. Subjects who have evidence or history of clinically significant allergic (except for untreated, asymptomatic, seasonal allergies at time of dosing), hematological, endocrine,pulmonary, gastrointestinal, cardiovascular, hepatic, psychiatric, or neurological disease. Exceptions to these criteria (eg, stable, mild joint disease) may be made following discussions with the Medical Monitor.
7. Subjects with a medical history of or who have a positive serology test for human immunodeficiency virus (HIV), hepatitis B virus surface antigen (HBsAg), or hepatitis C virus (HCV).
8. Subjects who have a history of drug or alcohol abuse or dependence within 18 months prior to Screening.
9. Subjects who have donated blood or blood components within the 4 weeks prior to Period 1 Check-in.
10. Subjects with laboratory values outside of the normal range for the local laboratory.
11. Subjects who have a sustained supine SBP >140 mmHg or <100 mm Hg or a DBP >95 mmHg at Screening or baseline.
12. Subjects who have a resting HR of <45 bpm or >100 bpm.
13. Subjects who have an abnormal Screening ECG indicating a second- or third-degree atrioventricular (AV) block, or 1 or more of the following: QRS interval >110 msec, QTc interval >450 msec, PR interval >240 msec, or any rhythm other than sinus rhythm, which is interpreted by the Investigator to be clinically significant.
14. Subjects who use or have used tobacco-containing products within the 6 months prior to Period 1 Check-in and throughout the study.
15. Subjects who have consumed alcohol-, caffeine-, or xanthine-containing products within 72 hours prior to Period 1 Check-in and throughout the study.
16. Subjects who test positive for drug(s) of abuse, alcohol, or cotinine at Screening or Check-in for any period.
17. Subjects who have concomitant medication usage of any nitrate, trazadone, ketoconozole, erythromycin, cimetidine, androgen replacement therapy and/or use of other prescription or over-the-counter drugs that are known to interfere with metabolism by CYP3A4.
18. Subjects who have used any drug that may prolong the QT/QTc interval within 30 days.
19. Subjects who have used a prescription drug or over-the-counter or herbal medication within 14 days
20. Subjects who are involved in the planning and/or conduct of the study.
21. Subjects who, for any reason, are deemed by the Investigator to be inappropriate for this study, including subjects who are unable to communicate or to cooperate with the Investigator.

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 57 (Actual)
Dates: Start 2008-10; Primary Completion 2009-01 (Actual); Study Completion 2009-01 (Actual)

PRIMARY OUTCOMES:
Time-matched change from baseline in QTcI that provides optimization of QT correction of heart rate as compared to fixed exponent approaches such as QTcB or QTcF. | 24 Hours

CONTACTS AND LOCATIONS:
Overall Officials: Chuck Bowden, M.D., Study Director — VIVUS LLC
Locations (1):
- Covance Phase 1 Clinical Unit, Madison, Wisconsin, United States